CLINICAL TRIAL: NCT07211074
Title: Optimal Positive End-Expiratory Pressure (PEEP) Level for Minimizing the Risk of Postoperative Atelectasis According to Lung Ultrasound Monitoring: A Retrospective Cohort Study
Brief Title: Optimal PEEP Level for Minimizing the Risk of Postoperative Atelectasis: A Retrospective Cohort Study Based on Lung Ultrasound Monitoring
Acronym: ULTRASVENT-1
Status: Completed | Type: Observational
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Other Study IDs: NMSC-03-25
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pulmonary Complications (PPCs); Postoperative Atelectasis; Lung Ultrasound
Keywords: Postoperative Atelectasis; Lung Ultrasound; Postoperative Desaturation; Postoperative Pulmonary Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ETT with PEEP ≤7 cm H₂O: This cohort consists of patients who underwent surgery with general anesthesia managed with an endotracheal tube (ETT) and a positive end-expiratory pressure (PEEP) of 7 cm H₂O or less. This group will include 250 patients in the final analysis
- ETT with PEEP ≥8 cm H₂O: This cohort consists of patients who underwent surgery with general anesthesia managed with an endotracheal tube (ETT) and a positive end-expiratory pressure (PEEP) of 8 cm H₂O or greater. This group will include 119 patients in the final analysis
- Laryngeal Mask: This cohort consists of patients who underwent surgery with general anesthesia managed with a laryngeal mask (LM) for airway protection. This group will include 81 patients in the final analysis

SUMMARY:
Background: After surgery with general anesthesia, it is common for parts of the lungs to collapse, a condition called atelectasis. This can lead to low blood oxygen levels and other lung complications. Doctors use a setting on the breathing machine called PEEP (Positive End-Expiratory Pressure) to help keep the lungs open, but the best level to use is still debated.

Purpose of the Study: The goal of this research is to find a PEEP level that minimizes the risk of lung collapse and low oxygen levels after surgery. The investigators will use lung ultrasound, a safe and non-invasive imaging method, to check the health of the lungs at the patient's bedside.

The investigators will not assign treatments; they will observe the outcomes based on the PEEP level chosen by the patient's anesthesiologist during routine care. A simplified ultrasound scan will be used to score the amount of lung collapse before and after surgery. The main outcomes will be the frequency of lung collapse and the frequency of low oxygen levels (defined as SpO₂ of 90% or less).

DETAILED DESCRIPTION:
Background and Rationale Postoperative pulmonary complications (PPCs) are a significant cause of morbidity and mortality, associated with a nearly 20% increase in lethality and prolonged hospital stays. The most common PPC is atelectasis, which can trigger more severe complications and develops in up to 90% of patients following the induction of general anesthesia. While computed tomography (CT) is the gold standard for diagnosing atelectasis, lung ultrasound (LUS) has emerged as a rapid, reliable, and validated bedside tool that is superior to standard chest radiography, with a high sensitivity (87.7%) and specificity (92.1%) compared to CT.

A key strategy for preventing atelectasis is the application of positive end-expiratory pressure (PEEP). While ventilation with zero PEEP is considered harmful, the optimal level remains controversial. Large randomized trials (e.g., PROVHILO, PROBESE) have not shown a benefit for universally high PEEP strategies (e.g., 12 cm H₂O) and have noted an increased risk of hemodynamic instability. This contrasts with other studies suggesting benefits from moderate or individualized PEEP levels. This study designed to address this gap by analyzing data to identify a PEEP threshold associated with minimal atelectasis and desaturation, using a simplified LUS monitoring protocol.

Study Objectives The primary objective of this study is to evaluate the effectiveness of a simplified LUS protocol for monitoring postoperative atelectasis and to determine a PEEP level associated with the minimum frequency and severity of atelectasis.

Specific study tasks include:

* To assess the frequency and severity of postoperative atelectasis in patients with different airway management strategies and PEEP levels.
* To determine an optimal PEEP threshold for minimizing the risk of atelectasis and desaturation using ROC analysis.
* To compare the rates of atelectasis and desaturation (SpO₂ ≤90%) between patient subgroups.
* To conduct a multifactorial analysis of risk factors for developing postoperative atelectasis and desaturation.
* To evaluate the prognostic value of the LUS score for predicting the risk of postoperative desaturation.

Study Design and Methodology This is a single-center, retrospective cohort study conducted at the National Medical and Surgical Center n.a. N.I. Pirogov. The level of PEEP not assigned by the protocol but determined by the attending anesthesiologist as part of routine clinical practice.

A simplified 2-zone LUS protocol will be used, focusing on the posterior-basal lung regions most susceptible to collapse. Lung aeration will be quantified using a 4-point scoring system (0-3), with 0 indicating normal aeration and 3 indicating major consolidation. Scans will be performed by one of three competent investigators before anesthesia and within the first hours after surgery, once the patient is fully awake.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical intervention under general anesthesia with mechanical ventilation.
* Airway protection managed with either an endotracheal tube or a laryngeal mask.
* A normal baseline ultrasound of the posterior-basal lung regions, corresponding to a score of 0 on the lung ultrasound scale.

Exclusion Criteria:

* Patients undergoing cardiac or thoracic surgery.
* Presence of a perioperatively identified pneumothorax.
* Inability to obtain adequate ultrasound visualization of the target lung zones.
* Presence of hydrothorax.
* Confirmed perioperative pulmonary aspiration.
* Presence of any pathological findings on the initial baseline ultrasound of the posterior-basal lung regions.
* Requirement for massive blood transfusion during the operation.
* Patients undergoing surgery on the diaphragm.
* Prolonged residual sedation lasting more than 2 hours post-operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 450 adult patients who underwent surgical procedures under general anesthesia with mechanical ventilation. Data will be collected from patients treated at the Department of Anesthesiology and Resuscitation of the National Medical and Surgical Center n.a. N.I. Pirogov.
  The cohort will be formed using a time-stratified randomization method to ensure a representative sample over the study period. All included patients will have a normal lung ultrasound before their procedure.
  The population will be divided based on the method of airway protection:
  * patients managed with an endotracheal tube (ETT).
  * patients managed with a laryngeal mask (LM).
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2025-09-22 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
Frequency of Postoperative Atelectasis | The ultrasound measurement is performed within the first few hours after the completion of the surgical procedure
  The measure assesses the presence of postoperative atelectasis, defined as a lung ultrasound (LUS) score greater than 0. The assessment is conducted using a simplified 2-zone LUS protocol, with aeration evaluated on a 4-point scale (from 0 for normal aeration to 3 for major consolidation). The outcome is the percentage of patients who develop any degree of atelectasis (LUS score > 0) following surgery

SECONDARY OUTCOMES:
Frequency of Postoperative Desaturation | Within the first few hours after completion of surgery
  The percentage of patients who experience an episode of clinically significant postoperative desaturation. This is defined as a peripheral oxygen saturation (SpO₂) of 90% or less. The measurement is recorded after the patient is fully awake and breathing spontaneously
Severity of Postoperative Atelectasis Measured by Lung Ultrasound Score | The final LUS score is measured within the first few hours after completion of surgery
  The overall severity of postoperative atelectasis, measured by the total score from the lung ultrasound (LUS) assessment. The score is a quantitative value from 0 to 6 (up to 3 points for each of the two lung zones). This outcome is analyzed as a continuous variable, comparing the median scores between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Teplykh, MD, Study Director — Pirogov National Medical and Surgical Center; Ivan Shcheparev, MD, PhD, Principal Investigator — Pirogov National Medical and Surgical Center
Locations (1):
- Pirogov National Medical and Surgical Cente, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 2 months after completion of the study
Access Criteria: upon the request

REFERENCES:
- [Background] Writing Committee for the PROBESE Collaborative Group of the PROtective VEntilation Network (PROVEnet) for the Clinical Trial Network of the European Society of Anaesthesiology; Bluth T, Serpa Neto A, Schultz MJ, Pelosi P, Gama de Abreu M; PROBESE Collaborative Group; Bluth T, Bobek I, Canet JC, Cinnella G, de Baerdemaeker L, Gama de Abreu M, Gregoretti C, Hedenstierna G, Hemmes SNT, Hiesmayr M, Hollmann MW, Jaber S, Laffey J, Licker MJ, Markstaller K, Matot I, Mills GH, Mulier JP, Pelosi P, Putensen C, Rossaint R, Schmitt J, Schultz MJ, Senturk M, Serpa Neto A, Severgnini P, Sprung J, Vidal Melo MF, Wrigge H. Effect of Intraoperative High Positive End-Expiratory Pressure (PEEP) With Recruitment Maneuvers vs Low PEEP on Postoperative Pulmonary Complications in Obese Patients: A Randomized Clinical Trial. JAMA. 2019 Jun 18;321(23):2292-2305. doi: 10.1001/jama.2019.7505. PMID 31157366
- [Background] Mazzinari G, Zampieri FG, Ball L, Campos NS, Bluth T, Hemmes SNT, Ferrando C, Librero J, Soro M, Pelosi P, Gama de Abreu M, Schultz MJ, Serpa Neto A; for REPEAT on behalf of the PROVHILO, iPROVE, and PROBESE investigators and the PROVE Network investigators. High Positive End-expiratory Pressure (PEEP) with Recruitment Maneuvers versus Low PEEP during General Anesthesia for Surgery: A Bayesian Individual Patient Data Meta-analysis of Three Randomized Clinical Trials. Anesthesiology. 2025 Jan 1;142(1):72-97. doi: 10.1097/ALN.0000000000005170. PMID 39042027
- [Background] Yoon HK, Kim BR, Yoon S, Jeong YH, Ku JH, Kim WH. The Effect of Ventilation with Individualized Positive End-Expiratory Pressure on Postoperative Atelectasis in Patients Undergoing Robot-Assisted Radical Prostatectomy: A Randomized Controlled Trial. J Clin Med. 2021 Feb 19;10(4):850. doi: 10.3390/jcm10040850. PMID 33669526
- [Background] Cho S, Oh HW, Choi MH, Lee HJ, Woo JH. Effects of Intraoperative Ventilation Strategy on Perioperative Atelectasis Assessed by Lung Ultrasonography in Patients Undergoing Open Abdominal Surgery: a Prospective Randomized Controlled Study. J Korean Med Sci. 2020 Oct 12;35(39):e327. doi: 10.3346/jkms.2020.35.e327. PMID 33045769
- [Background] Young CC, Harris EM, Vacchiano C, Bodnar S, Bukowy B, Elliott RRD, Migliarese J, Ragains C, Trethewey B, Woodward A, Gama de Abreu M, Girard M, Futier E, Mulier JP, Pelosi P, Sprung J. Lung-protective ventilation for the surgical patient: international expert panel-based consensus recommendations. Br J Anaesth. 2019 Dec;123(6):898-913. doi: 10.1016/j.bja.2019.08.017. Epub 2019 Oct 3. PMID 31587835
- [Background] Ma J, Sun M, Song F, Wang A, Tian X, Wu Y, Wang L, Zhao Q, Liu B, Wang S, Qiu Y, Hou H, Deng L. Effect of ultrasound-guided individualized positive end-expiratory pressure on the severity of postoperative atelectasis in elderly patients: a randomized controlled study. Sci Rep. 2024 Nov 15;14(1):28128. doi: 10.1038/s41598-024-79105-8. PMID 39548165
- [Background] Liao B, Liao W, Yin S, Liu S, Wu X. Effect of ultrasound-guided lung recruitment to reduce pulmonary atelectasis after non-cardiac surgery under general anesthesia: a systematic review and meta-analysis of randomized controlled trials. Perioper Med (Lond). 2024 Mar 27;13(1):23. doi: 10.1186/s13741-024-00379-7. PMID 38539248
- [Background] Wu XZ, Xia HM, Zhang P, Li L, Hu QH, Guo SP, Li TY. Effects of ultrasound-guided alveolar recruitment manoeuvres compared with sustained inflation or no recruitment manoeuvres on atelectasis in laparoscopic gynaecological surgery as assessed by ultrasonography: a randomized clinical trial. BMC Anesthesiol. 2022 Aug 16;22(1):261. doi: 10.1186/s12871-022-01798-z. PMID 35974310
- See also: Official website of the Pirogov National Medical and Surgical Center — https://www.pirogov-center.ru/english/about/